CLINICAL TRIAL: NCT06457763
Title: Comparison of Ultrasound and Classical Method for Left Double Lumen Tube Selection in One-Lung Ventilation: A Randomised Controlled Study
Brief Title: Left Double Lumen Tube Selection
Status: Completed | Type: Observational
Sponsor: Marmara University (Other)
Responsible Party: Principal Investigator, Meliha Orhon, Assistant professor, Marmara University
Other Study IDs: 09.2022.755
Record Dates: First submitted 2024-05-29; First posted 2024-06-13 (Actual); Last update posted 2024-06-25 (Actual); Status verified 2024-06

CONDITIONS: One-Lung Ventilation; Thoracic Surgery
Keywords: Ultrasound; Double lumen tube; Postoperative complication
MeSH Terms: conditions — Postoperative Complications

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 6 Months
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Ultrasound: While the patients were in the supine position on the operating room table, the external tracheal diameter, measured just above the sternoclavicular junction, was measured by ultrasound. Appropriately sized tube size was selected in accordance with previous studies and cadaver studies.
- conventional: For female patients, a 37 fr left double lumen tube was chosen for patients taller than 160 cm, and a 35 fr left double lumen tube was chosen for patients shorter than 160 cm. For male patients, a 41 fr left double lumen tube was selected for patients taller than 170 cm and a 39 fr tube was chosen for men shorter than 170 cm.

SUMMARY:
The aim of this study was to determine the accuracy and practicality of ultrasound in the selection of double lumen tube and whether the complications that may occur intraoperatively and postoperatively can be reduced.

Patients aged 18-75 years with ASA 1-2-3 who give informed consent for left double lumen tube placement for single lung ventilation will be included in this study. Patients with a history of previous difficult intubation, head and neck surgery and radiotherapy, class 3-4 in the Colmark-Lehane classification by the thoracic anaesthetist who will perform the intubation, and patients with previously known hoarseness and chronic cough will not be included in the study. Patients who accept the study will be randomly assigned to one of the anaesthesia groups including ultrasound group (Group 1) and classical method (Group 2).

Randomisation will be in a 1:1 ratio and will be done by closed envelope method.

DETAILED DESCRIPTION:
The aim of this study was to determine the accuracy and practicality of ultrasound in the selection of double lumen tube and whether the complications that may occur intraoperatively and postoperatively can be reduced.

In thoracic surgery, single lung ventilation is one of the most challenging airway and ventilation methods for anaesthetists. Bronchial blockers and double lumen tubes are the tools used to isolate the lung in single lung ventilation and double lumen tubes are used more frequently. Size is important when choosing a double lumen tube. There is no definite rule when choosing the tube size. When selecting the size of the double lumen tube, there is a classical method selected according to the gender and height of the patient. However, due to anatomical differences between individuals; inappropriate tube sizes may be selected and this may lead to consequences such as tracheabronchial injury and insufficient deflation of the lungs.

The use of ultrasound can provide rapid assessment of airway anatomy in the operating theatre, intensive care unit and emergency department. Ultrasound is a suitable tool for the evaluation of the subglottic airway confirmed by computed tomography. The use of ultrasound requires less training and the patient does not need to be fully immobilised and sedated. There is a correlation between the diameter of the external trachea measured by ultrasound just above the sternoclavicular junction and the diameter of the left main bronchus measured by computed tomography scan.

Patients aged 18-75 years with ASA 1-2-3 who give informed consent for left double lumen tube placement for single lung ventilation will be included in this study. Patients with a history of previous difficult intubation, head and neck surgery and radiotherapy, class 3-4 in the Colmark-Lehane classification by the thoracic anaesthetist who will perform the intubation, and patients with previously known hoarseness and chronic cough will not be included in the study. Patients who accept the study will be randomly assigned to one of the anaesthesia groups including ultrasound group (Group 1) and classical method (Group 2).

Randomisation will be in a 1:1 ratio and will be done by closed envelope method. A paper with the name of one of the two groups will be placed in the envelopes beforehand and the envelopes will be closed and mixed. For each patient, a closed envelope will be drawn randomly before the procedure and the procedures will be performed according to the group indicated on the paper.

Intraoperative anaesthesia management Before induction of anaesthesia, the patients in this group will be placed in the supine position with the head in slight extension and the outer diameter of the trachea will be measured with a linear probe 0.5 cm above the sternoclavicular joint by placing the ultrasound transverse and the patient will be intubated by selecting a left double lumen tube suitable for this measurement.

In the classical method group (Group2), 37 fr left double lumen tube was selected for female patients taller than 160 cm and 35 fr left double lumen tube was selected for patients shorter than 160 cm. For male patients, a 41 fr left double lumen tube was selected for patients taller than 170 cm and a 39 fr tube was selected for men shorter than 170 cm.

Anaesthesia induction was performed with propofol (2 mg/kg), remifentanil 1mcg/kg, and rocuronium 0.6 mg/kg under standard monitoring (ECG, non-invasive blood pressure, and finger prick oxygen saturation). In both groups of patients, after direct laryngoscopy and visualisation of the vocal cords, the tip of the left double lumen tube was rotated 90 degrees counterclockwise past the vocal cords and pushed until resistance was felt. The depth of the left double lumen tube was determined as 12+ patient height (cm)/10 cm from the tooth level and then the location of the tube was confirmed with a fibreoptic bronchoscope.

ELIGIBILITY:
Inclusion Criteria:

* Patients who will place a left double lumen tube to perform one lung ventilation
* Between the ages of 18-75
* ASA 1-2-3 patients

Exclusion Criteria:

* Patients with a previous history of difficult intubation
* Patients who have previously undergone head and neck surgery or received radiotherapy
* Patients with a Cormark-Lehane classification of 3-4 by the thoracic anaesthetist performing intubation,
* Patients with previous cough and sore throat

Ages: 18 Years to 75 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: Patients aged 18-75 years, ASA 1-2-3 and giving informed consent
Sampling Method: Probability Sample
Enrollment: 70 (Actual)
Dates: Start 2023-08-01 (Actual); Primary Completion 2023-09-01 (Actual); Study Completion 2024-05-29 (Actual)

PRIMARY OUTCOMES:
postoperative cough and sore throat | postoperative first at 24 hours
  Zero: No sore throat; 1: Mild, sore throat only when swallowing; 2: Moderate, persistent sore throat, aggravated when swallowing; 3: Severe, throat pain affecting the patient's eating, and analgesic drugs were needed

CONTACTS AND LOCATIONS:
Locations (1):
- Marmara University, Istanbul, Maltepe, Turkey (Türkiye)